CLINICAL TRIAL: NCT01055353
Title: Evaluation of Target Organs Damage in Hypertensive Patients Followed in General Practice With no Known Cardiovascular (CV) or Renal Disease, Stratified According to Blood Pressure Control
Brief Title: Evaluation of Target Organs Damage in Hypertensive Patients
Acronym: PreVENT-A GP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC CD, AstraZeneca
Other Study IDs: NIS-CFR-DUM-2009/2
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Target Organs Damage; Hypertensive; no Known Cardiovascular; no Known Renal Disease
Keywords: Target organs damage; hypertensive patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of target organs damage in hypertensive patients with no known cardiovascular (CV) or renal disease, stratified according to level of blood pressure control

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of essential hypertension (treated or untreated); HT not discovered on the day of the consultation; no documented clinical cardiovascular or renal disease.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First 2 consecutive adults with hypertension, with no known cardiovascular (CV) or renal disease, seen by general practitioner
Sampling Method: Probability Sample
Enrollment: 1857 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the frequency of evaluation of preclinical target organs damage in hypertensive patients with no known cardiovascular or renal disease, by taking blood pressure (controlled or uncontrolled HT*) into account | once / 1 Year

SECONDARY OUTCOMES:
To describe the patient profile (socio-demographic, risk factors, comorbidities, global CV risk level estimated by the doctor and calculated retrospectively [according to ESH 2007]) associated with screening for target organs damage
To describe the modalities of patient follow-up and management
To compare the frequency of evaluation of target organs damage as a function of the modalities of management of CV risk factors at the time of the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Piedbois, Study Director — AstraZeneca
Locations (905):
- France (905):
  - Research Site, Abbaretz
  - Research Site, Achenheim
  - Research Site, Achères
  - Research Site, Achicourt
  - Research Site, Agde
  - Research Site, Aigurande
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Ajaccio
  - Research Site, Albertville
  - Research Site, Albi
  - Research Site, Alès
  - Research Site, Allaire
  - Research Site, Alligny-Cosne
  - Research Site, Allouagne
  - Research Site, Ambrières-les-Vallées
  - Research Site, Amiens
  - Research Site, Amphion-les-Bains
  - Research Site, Amplepuis
  - Research Site, Andance
  - Research Site, Andeville
  - Research Site, Annecy
  - Research Site, Annecy-le-Vieux
  - Research Site, Annonay
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Arbois
  - Research Site, Arc-et-Senans
  - Research Site, Arcachon
  - Research Site, Arches
  - Research Site, Argenteuil
  - Research Site, Arles
  - Research Site, Arras
  - Research Site, Ars
  - Research Site, Art-sur-Meurthe
  - Research Site, Artannes-sur-Indre
  - Research Site, Arudy
  - Research Site, Asnières-sur-Seine
  - Research Site, Athies
  - Research Site, Aubagne
  - Research Site, Aubervilliers
  - Research Site, Aubière
  - Research Site, Auby
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Auchy-les-Mines
  - Research Site, Audincourt
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aumale
  - Research Site, Aumont-Aubrac
  - Research Site, Autun
  - Research Site, Auxerre
  - Research Site, Avesnes-le-Sec
  - Research Site, Avignon
  - Research Site, Avoine
  - Research Site, Avrillé
  - Research Site, Badonviller
  - Research Site, Bagneux
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baignes Ste Radegonde
  - Research Site, Baisieux
  - Research Site, Balaruc-les-Bains
  - Research Site, Banyuls de la Marenda
  - Research Site, Barberaz
  - Research Site, Barbezieux-Saint-Hilaire
  - Research Site, Bassussarry
  - Research Site, Bayonne
  - Research Site, Bâgé-le-Châtel
  - Research Site, Beaulieu
  - Research Site, Beaumesnil
  - Research Site, Beaumont
  - Research Site, Beaumont-en-Véron
  - Research Site, Beaumont-sur-Lèze
  - Research Site, Beautor
  - Research Site, Beauvais
  - Research Site, Belleville-sur-Meuse
  - Research Site, Benfeld
  - Research Site, Benquet
  - Research Site, Bergerac
  - Research Site, Bergholtz
  - Research Site, Bersée
  - Research Site, Bertrichamps
  - Research Site, Bessines
  - Research Site, Beynes
  - Research Site, Bélâbre
  - Research Site, Bérat
  - Research Site, Bétaille
  - Research Site, Béville-le-Comte
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Biganos
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blanquefort
  - Research Site, Bohars
  - Research Site, Bois-Colombes
  - Research Site, Boisset
  - Research Site, Bondues
  - Research Site, Bondy
  - Research Site, Bordeaux
  - Research Site, Bort-les-Orgues
  - Research Site, Bouc-Bel-Air
  - Research Site, Boujan-sur-Libron
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourbriac
  - Research Site, Bourg-Achard
  - Research Site, Bourg-Argental
  - Research Site, Bourg-la-Reine
  - Research Site, Bourg-lès-Valence
  - Research Site, Bourges
  - Research Site, Bousbecque
  - Research Site, Boussay
  - Research Site, Bousse
  - Research Site, Bozel
  - Research Site, Braine
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Bretignolles-sur-Mer
  - Research Site, Breuil-le-Sec
  - Research Site, Brignais
  - Research Site, Brignoud
  - Research Site, Briollay
  - Research Site, Brion-près-Thouet
  - Research Site, Broût-Vernet
  - Research Site, Bruère-Allichamps
  - Research Site, Bubry
  - Research Site, Bulgnéville
  - Research Site, Bulles
  - Research Site, Cabanac-et-Villagrains
  - Research Site, Callac de Bretagne
  - Research Site, Caluire-et-Cuire
  - Research Site, Camblanes
  - Research Site, Cambrai
  - Research Site, Camors
  - Research Site, Campbon
  - Research Site, Canet-Plage
  - Research Site, Canéjan
  - Research Site, Cannes
  - Research Site, Cany-Barville
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Cappelle-en-Pévèle
  - Research Site, Carantec
  - Research Site, Carbon-Blanc
  - Research Site, Carcassonne
  - Research Site, Carentan
  - Research Site, Carnon-Plage
  - Research Site, Carpentras
  - Research Site, Carpiquet
  - Research Site, Carresse-Cassaber
  - Research Site, Carrières-sur-Seine
  - Research Site, Carros
  - Research Site, Cavaillon
  - Research Site, Celles-sur-Plaine
  - Research Site, Cerizay
  - Research Site, Cénac
  - Research Site, Cérilly
  - Research Site, Chaleins
  - Research Site, Chamalières
  - Research Site, Chambéry
  - Research Site, Chambray-lès-Tours
  - Research Site, Chamonix
  - Research Site, Champagnole
  - Research Site, Champcueil
  - Research Site, Champigneulles
  - Research Site, Champigny-sur-Marne
  - Research Site, Chanac
  - Research Site, Chantilly
  - Research Site, Chantonnay
  - Research Site, Charleville-Mézières
  - Research Site, Charmes
  - Research Site, Charmoy
  - Research Site, Chasseneuil-du-Poitou
  - Research Site, Chauvigny
  - Research Site, Châbons
  - Research Site, Château-Chinon(Ville)
  - Research Site, Château-Thierry
  - Research Site, Châteaubriant
  - Research Site, Châteauneuf-en-Thymerais
  - Research Site, Châteauneuf-sur-Cher
  - Research Site, Châtellerault
  - Research Site, Châtenay-Malabry
  - Research Site, Châtillon-Coligny
  - Research Site, Châtillon-sur-Colmont
  - Research Site, Cherbourg Octeville
  - Research Site, Cherves-Richemont
  - Research Site, Chinon
  - Research Site, Ciboure
  - Research Site, Cinq-Mars-la-Pile
  - Research Site, Ciry-le-Noble
  - Research Site, Clairac
  - Research Site, Clary
  - Research Site, Clermont-Ferrand
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Cluny
  - Research Site, Cognac
  - Research Site, Collioure
  - Research Site, Colomars
  - Research Site, Colombes
  - Research Site, Colomiers
  - Research Site, Combrit
  - Research Site, Commentry
  - Research Site, Conches-en-Ouche
  - Research Site, Condrieu
  - Research Site, Connaux
  - Research Site, Corbehem
  - Research Site, Corbeil-Essonnes
  - Research Site, Corcieux
  - Research Site, Corseul
  - Research Site, Coudekerque-Branche
  - Research Site, Couhé
  - Research Site, Courbevoie
  - Research Site, Courcy
  - Research Site, Cournon-d'Auvergne
  - Research Site, Courpière
  - Research Site, Courrières
  - Research Site, Coursan
  - Research Site, Courthézon
  - Research Site, Coutances
  - Research Site, Coutouvre
  - Research Site, Coye-la-Forêt
  - Research Site, Cran-Gevrier
  - Research Site, Creil
  - Research Site, Crécy-sur-Serre
  - Research Site, Créteil
  - Research Site, Crévic
  - Research Site, Criquetot-l'Esneval
  - Research Site, Croissy-sur-Seine
  - Research Site, Croix
  - Research Site, Cubjac
  - Research Site, Cugand
  - Research Site, Cunlhat
  - Research Site, Dainville
  - Research Site, Dambach-la-Ville
  - Research Site, Deauville
  - Research Site, Dieppe
  - Research Site, Dieulouard
  - Research Site, Dieuze
  - Research Site, Dijon
  - Research Site, Dinard
  - Research Site, Dinsheim-sur-Bruche
  - Research Site, Dole
  - Research Site, Domfront
  - Research Site, Dornes
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Elna
  - Research Site, Enghien-les-Bains
  - Research Site, Entraygues-sur-Truyère
  - Research Site, Eragny Sur Oise
  - Research Site, Ermont
  - Research Site, Escaudain
  - Research Site, Esquerdes
  - Research Site, Estaing
  - Research Site, Eyguières
  - Research Site, Échenoz-la-Méline
  - Research Site, Échirolles
  - Research Site, Épernon
  - Research Site, Épierre
  - Research Site, Épinal
  - Research Site, Épinay-sur-Seine
  - Research Site, Épron
  - Research Site, Étalondes
  - Research Site, Étretat
  - Research Site, Étupes
  - Research Site, Évin-Malmaison
  - Research Site, Évron
  - Research Site, Ézy-sur-Eure
  - Research Site, Fabrezan
  - Research Site, Faches-Thumesnil
  - Research Site, Fameck
  - Research Site, Faverges
  - Research Site, Fegersheim
  - Research Site, Felletin
  - Research Site, Fère-en-Tardenois
  - Research Site, Fécamp
  - Research Site, Félines
  - Research Site, Firmi
  - Research Site, Firminy
  - Research Site, Fitilieu
  - Research Site, Fitz-James
  - Research Site, Flers
  - Research Site, Fleurance
  - Research Site, Florensac
  - Research Site, Folembray
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Fontès
  - Research Site, Fos-sur-Mer
  - Research Site, Fosses
  - Research Site, Fouras
  - Research Site, Fourneaux
  - Research Site, Franconville
  - Research Site, Frasne
  - Research Site, Fresnes-sur-Escaut
  - Research Site, Fréjus
  - Research Site, Froberville
  - Research Site, Fromentine
  - Research Site, Frontenex
  - Research Site, Frotey-lès-Vesoul
  - Research Site, Fyé
  - Research Site, Gaillefontaine
  - Research Site, Gallardon
  - Research Site, Gardonne
  - Research Site, Gelles
  - Research Site, Gelos
  - Research Site, Gennevilliers
  - Research Site, Gentilly
  - Research Site, Golbey
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gorcy
  - Research Site, Grandris
  - Research Site, Grane
  - Research Site, Granville
  - Research Site, Grasse
  - Research Site, Grenoble
  - Research Site, Gréasque
  - Research Site, Guerville
  - Research Site, Guérande
  - Research Site, Guidel
  - Research Site, Guignicourt
  - Research Site, Guiscriff
  - Research Site, Guise
  - Research Site, Hagondange
  - Research Site, Hanvec
  - Research Site, Harnes
  - Research Site, Hendaye
  - Research Site, Hénin-Beaumont
  - Research Site, Horbourg-Wihr
  - Research Site, Houilles
  - Research Site, Hundling
  - Research Site, Hyères
  - Research Site, Isbergues
  - Research Site, Isle
  - Research Site, Issy-les-Moulineaux
  - Research Site, Ivry-sur-Seine
  - Research Site, Jacou
  - Research Site, Jardin
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jassans-Riottier
  - Research Site, Jeumont
  - Research Site, Joinville-le-Pont
  - Research Site, Jonquières
  - Research Site, Jonquières-Saint-Vincent
  - Research Site, Jouars-Pontchartrain
  - Research Site, Joué-lès-Tours
  - Research Site, Jugon-les-Lacs
  - Research Site, Jujurieux
  - Research Site, Jussey
  - Research Site, L'Haÿ-les-Roses
  - Research Site, La Bernerie-en-Retz
  - Research Site, La Bouilladisse
  - Research Site, La Chapelaude
  - Research Site, La Couronne
  - Research Site, La Crau
  - Research Site, La Fère
  - Research Site, La Fouillade
  - Research Site, La Francheville
  - Research Site, La Frette-sur-Seine
  - Research Site, La Garde
  - Research Site, La Garnache
  - Research Site, La Grand-Combe
  - Research Site, La Haye-Pesnel
  - Research Site, La Madeleine
  - Research Site, La Mézière
  - Research Site, La Mothe-Saint-Héray
  - Research Site, La Motte-Servolex
  - Research Site, La Mulatière
  - Research Site, La Neuville-Roy
  - Research Site, La Queue-en-Brie
  - Research Site, La Réole
  - Research Site, La Ricamarie
  - Research Site, La Riche
  - Research Site, La Roche-sur-Foron
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Tour-de-Salvagny
  - Research Site, La Tranche-sur-Mer
  - Research Site, La Trimouille
  - Research Site, La Trinité-sur-Mer
  - Research Site, La Turballe
  - Research Site, La Varenne-Saint-Hilaire
  - Research Site, Labastidette
  - Research Site, Lacaune
  - Research Site, Laissac
  - Research Site, Lamagistère
  - Research Site, Lamballe
  - Research Site, Lambersart
  - Research Site, Lamorlaye
  - Research Site, Lamotte-Beuvron
  - Research Site, Lampertheim
  - Research Site, Landerneau
  - Research Site, Landes
  - Research Site, Landouge
  - Research Site, Lanester
  - Research Site, Langoiran
  - Research Site, Langres
  - Research Site, Lanildut
  - Research Site, Lanmeur
  - Research Site, Lannion
  - Research Site, Largentière
  - Research Site, Lathus-Saint-Rémy
  - Research Site, Latresne
  - Research Site, Lavit
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Bourget-du-Lac
  - Research Site, Le Bouscat
  - Research Site, Le Cannet
  - Research Site, Le Château-d’Oléron
  - Research Site, Le Chesnay
  - Research Site, Le Clion-sur-Mer
  - Research Site, Le Fenouiller
  - Research Site, Le Golfe Juan
  - Research Site, Le Grand-Quevilly
  - Research Site, Le Havre
  - Research Site, Le Mans
  - Research Site, Le Mée-sur-Seine
  - Research Site, Le Mêle-sur-Sarthe
  - Research Site, Le Plessis-Robinson
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Pont-de-Beauvoisin
  - Research Site, Le Rouret
  - Research Site, Le Soler
  - Research Site, Le Teil
  - Research Site, Le Tignet
  - Research Site, Le Touquet-Paris-Plage
  - Research Site, Le Tréport
  - Research Site, Le Val D Albian
  - Research Site, Lens
  - Research Site, Les Forges
  - Research Site, Les Issambres
  - Research Site, Les Mées
  - Research Site, Les Mureaux
  - Research Site, Les Pennes-Mirabeau
  - Research Site, Les Ponts-de-Cé
  - Research Site, Les Sables-d'Olonne
  - Research Site, Levallois-Perret
  - Research Site, Lezoux
  - Research Site, Lévignac
  - Research Site, Lézignan-Corbières
  - Research Site, Liffol-le-Grand
  - Research Site, Liffré
  - Research Site, Lignières-Châtelain
  - Research Site, Ligny-en-Barrois
  - Research Site, Lille
  - Research Site, Limeil-Brévannes
  - Research Site, Limeray
  - Research Site, Limoux
  - Research Site, Lognes
  - Research Site, Loison-sous-Lens
  - Research Site, Lombez
  - Research Site, Lomme
  - Research Site, Longages
  - Research Site, Longueau
  - Research Site, Longué-Jumelles
  - Research Site, Loperhet
  - Research Site, Lorgues
  - Research Site, Lorient
  - Research Site, Lormont
  - Research Site, Louannec
  - Research Site, Loudun
  - Research Site, Lourdes
  - Research Site, Louveciennes
  - Research Site, Luçay-le-Mâle
  - Research Site, Lunéville
  - Research Site, Lurcy-Lévis
  - Research Site, Lyon
  - Research Site, Lys-lez-Lannoy
  - Research Site, Mably
  - Research Site, Magland
  - Research Site, Maintenon
  - Research Site, Maisons-Alfort
  - Research Site, Malissard
  - Research Site, Mamers
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Mantes-la-Ville
  - Research Site, Marange-Silvange
  - Research Site, Marcillac-la-Croisille
  - Research Site, Marcilly-en-Villette
  - Research Site, Marckolsheim
  - Research Site, Marcq-en-Barœul
  - Research Site, Marignane
  - Research Site, Marles-les-Mines
  - Research Site, Marly
  - Research Site, Marquion
  - Research Site, Marsac-en-Livradois
  - Research Site, Marseille
  - Research Site, Martignas-sur-Jalle
  - Research Site, Marvejols
  - Research Site, Masnières
  - Research Site, Masseret
  - Research Site, Mauguio
  - Research Site, Maule
  - Research Site, Mauléon-Licharre
  - Research Site, Maxéville
  - Research Site, Mayenne
  - Research Site, Mayet
  - Research Site, Mazan
  - Research Site, Meaux
  - Research Site, Meistratzheim
  - Research Site, Mesvres
  - Research Site, Metz
  - Research Site, Meulan-en-Yvelines
  - Research Site, Meximieux
  - Research Site, Mezel
  - Research Site, Mezzavia
  - Research Site, Méjannes-lès-Alès
  - Research Site, Méounes-lès-Montrieux
  - Research Site, Mérignac
  - Research Site, Mézidon-Canon
  - Research Site, Mimet
  - Research Site, Miramas
  - Research Site, Mirande
  - Research Site, Miribel-les-Échelles
  - Research Site, Mittersheim
  - Research Site, Moissac
  - Research Site, Moncé-en-Belin
  - Research Site, Moncrabeau
  - Research Site, Monpazier
  - Research Site, Montauban
  - Research Site, Montbrison
  - Research Site, Montceau-les-Mines
  - Research Site, Montcy-Notre-Dame
  - Research Site, Montendre
  - Research Site, Montesson
  - Research Site, Montélimar
  - Research Site, Montfavet
  - Research Site, Montfort-en-Chalosse
  - Research Site, Montguyon
  - Research Site, Montlouis-sur-Loire
  - Research Site, Montluçon
  - Research Site, Montmélian
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montrevel-en-Bresse
  - Research Site, Montrond-le-Château
  - Research Site, Montrond-les-Bains
  - Research Site, Montrouge
  - Research Site, Monts-sur-Guesnes
  - Research Site, Morestel
  - Research Site, Morhange
  - Research Site, Morteau
  - Research Site, Mouchin
  - Research Site, Mougins
  - Research Site, Moulay
  - Research Site, Moussey
  - Research Site, Moussy-le-Neuf
  - Research Site, Moustiers Ste Marie
  - Research Site, Moutiers Tarentaise
  - Research Site, Moutiers-les-Mauxfaits
  - Research Site, Mouvaux
  - Research Site, Mouy
  - Research Site, Moyeuvre-Grande
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Nasbinals
  - Research Site, Neauphle-le-Château
  - Research Site, Neufchâtel-en-Saosnois
  - Research Site, Neufchef
  - Research Site, Neuville-en-Ferrain
  - Research Site, Neuvy-sur-Barangeon
  - Research Site, Nevers
  - Research Site, Nexon
  - Research Site, Nègrepelisse
  - Research Site, Nérac
  - Research Site, Néré
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-le-Phaye
  - Research Site, Nogent-le-Rotrou
  - Research Site, Nogent-sur-Oise
  - Research Site, Noisiel
  - Research Site, Noisy-le-Grand
  - Research Site, Nordausques
  - Research Site, Notre-Dame-d'Oé
  - Research Site, Notre-Dame-de-Gravenchon
  - Research Site, Nouzonville
  - Research Site, Noyant-la-Gravoyère
  - Research Site, Noyen-sur-Sarthe
  - Research Site, Noyon
  - Research Site, Ohlungen
  - Research Site, Oignies
  - Research Site, Oisemont
  - Research Site, Ollioules
  - Research Site, Orange
  - Research Site, Orbec
  - Research Site, Orcines
  - Research Site, Origny Ste Benoite
  - Research Site, Ormes
  - Research Site, Orry-la-Ville
  - Research Site, Orthez
  - Research Site, Orvault
  - Research Site, Ouroux-sur-Saône
  - Research Site, Oyonnax
  - Research Site, Pagny-sur-Moselle
  - Research Site, Paillencourt
  - Research Site, Pantin
  - Research Site, Paris
  - Research Site, Paron
  - Research Site, Pau
  - Research Site, Pauillac
  - Research Site, Pernes-les-Fontaines
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Peyrestortes
  - Research Site, Peyruis
  - Research Site, Pfaffenhoffen
  - Research Site, Pierrepont-sur-Avre
  - Research Site, Pleaux
  - Research Site, Ploemeur
  - Research Site, Plourhan
  - Research Site, Plouzané
  - Research Site, Poissy
  - Research Site, Pont-Aven
  - Research Site, Pont-Croix
  - Research Site, Pont-de-Buis-lès-Quimerch
  - Research Site, Pont-de-l'Arche
  - Research Site, Pontailler-sur-Saône
  - Research Site, Pontault-Combault
  - Research Site, Pontivy
  - Research Site, Port Leucate
  - Research Site, Pouzay
  - Research Site, Pradines
  - Research Site, Préchac
  - Research Site, Prignac-et-Marcamps
  - Research Site, Pulnoy
  - Research Site, Puteaux
  - Research Site, Quessoy
  - Research Site, Questembert
  - Research Site, Quimper
  - Research Site, Quincy-sous-Sénart
  - Research Site, Quincy-Voisins
  - Research Site, Raismes
  - Research Site, Rambervillers
  - Research Site, Rauzan
  - Research Site, Râches
  - Research Site, Rânes
  - Research Site, Redon
  - Research Site, Reichshoffen
  - Research Site, Reiningue
  - Research Site, Remiremont
  - Research Site, Richardménil
  - Research Site, Richemont
  - Research Site, Rieupeyroux
  - Research Site, Rieux
  - Research Site, Rigney
  - Research Site, Rilhac-Rancon
  - Research Site, Ris-Orangis
  - Research Site, Rivery
  - Research Site, Roanne
  - Research Site, Robion
  - Research Site, Roche-la-Molière
  - Research Site, Rodez
  - Research Site, Rodilhan
  - Research Site, Rognes
  - Research Site, Rohrbach-lès-Bitche
  - Research Site, Rohrwiller
  - Research Site, Roisel
  - Research Site, Romagné
  - Research Site, Rombas
  - Research Site, Roncq
  - Research Site, Roquebrune-Cap-Martin
  - Research Site, Roquefort-sur-Soulzon
  - Research Site, Rosny-sous-Bois
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rousson
  - Research Site, Routot
  - Research Site, Rueil-Malmaison
  - Research Site, Ruffec
  - Research Site, Rully
  - Research Site, Sains-du-Nord
  - Research Site, Saint Georges Baillargeaux
  - Research Site, Saint Marc Sur Mer
  - Research Site, Saint Maximin La Ste Baume
  - Research Site, Saint-Affrique
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-André-des-Eaux
  - Research Site, Saint-Anthème
  - Research Site, Saint-Astier
  - Research Site, Saint-Aubin-des-Châteaux
  - Research Site, Saint-Barthélemy-de-Vals
  - Research Site, Saint-Barthélémy
  - Research Site, Saint-Benoît
  - Research Site, Saint-Bonnet-sur-Gironde
  - Research Site, Saint-Brevin-les-Pins
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Cézaire-sur-Siagne
  - Research Site, Saint-Chamond
  - Research Site, Saint-Cloud
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-lès-Bourg
  - Research Site, Saint-Dizier
  - Research Site, Saint-Donat-sur-l'Herbasse
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Etienne-de-Tulmont
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Étienne-lès-Remiremont
  - Research Site, Saint-Félix-de-Lodez
  - Research Site, Saint-Gaudens
  - Research Site, Saint-Genest-Malifaux
  - Research Site, Saint-Genis-les-Ollières
  - Research Site, Saint-Georges-de-Reneins
  - Research Site, Saint-Georges-des-Groseillers
  - Research Site, Saint-Georges-du-Bois
  - Research Site, Saint-Georges-sur-Baulche
  - Research Site, Saint-Germain-les-Belles
  - Research Site, Saint-Germainmont
  - Research Site, Saint-Gervais-d'Auvergne
  - Research Site, Saint-Girons
  - Research Site, Saint-Guénolé
  - Research Site, Saint-Hilaire-des-Loges
  - Research Site, Saint-Hilaire-lez-Cambrai
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-du-Gard
  - Research Site, Saint-Jean-Pied-de-Port
  - Research Site, Saint-Julien-de-Civry
  - Research Site, Saint-Just-Chaleyssin
  - Research Site, Saint-Just-en-Chaussée
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Lon-les-Mines
  - Research Site, Saint-Louis
  - Research Site, Saint-Mamert-du-Gard
  - Research Site, Saint-Marcellin
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-du-Var
  - Research Site, Saint-Martin-le-Beau
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice-des-Lions
  - Research Site, Saint-Max
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Nicolas-de-Port
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Palais-sur-Mer
  - Research Site, Saint-Paul-en-Chablais
  - Research Site, Saint-Philbert-de-Bouaine
  - Research Site, Saint-Pierre-d'Albigny
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-en-Val
  - Research Site, Saint-Pierre-le-Moûtier
  - Research Site, Saint-Porchaire
  - Research Site, Saint-Pourçain-sur-Sioule
  - Research Site, Saint-Priest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Quentin-la-Poterie
  - Research Site, Saint-Rambert-d'Albon
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-Sauveur-dAunis
  - Research Site, Saint-Sauveur-le-Vicomte
  - Research Site, Saint-Savournin
  - Research Site, Salbris
  - Research Site, Salernes
  - Research Site, Sanary-sur-Mer
  - Research Site, Sannois
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Saulnot
  - Research Site, Sault-lès-Rethel
  - Research Site, Saulxures-sur-Moselotte
  - Research Site, Sautron
  - Research Site, Sauveterre-de-Rouergue
  - Research Site, Saverne
  - Research Site, Savigné-l'Évêque
  - Research Site, Savonnières
  - Research Site, Sceaux
  - Research Site, Schiltigheim
  - Research Site, Schweighouse-sur-Moder
  - Research Site, Sedan
  - Research Site, Segonzac
  - Research Site, Segré
  - Research Site, Seichamps
  - Research Site, Sens
  - Research Site, Seraincourt
  - Research Site, Sers
  - Research Site, Sevran
  - Research Site, Sète
  - Research Site, Sélestat
  - Research Site, Sérignan
  - Research Site, Sigean
  - Research Site, Simiane-Collongue
  - Research Site, Six-Fours-les-Plages
  - Research Site, Socx
  - Research Site, Soissons
  - Research Site, Solre-le-Château
  - Research Site, Sonchamp
  - Research Site, Soucy
  - Research Site, Soufflenheim
  - Research Site, Souillac
  - Research Site, Soyaux
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Ste Bazeille
  - Research Site, Ste Florine
  - Research Site, Ste Fortunade
  - Research Site, Ste Menehould
  - Research Site, Ste Suzanne
  - Research Site, Strasbourg
  - Research Site, Sucy-en-Brie
  - Research Site, Suresnes
  - Research Site, Tarascon
  - Research Site, Tarascon-sur-Ariège
  - Research Site, Tassin-la-Demi-Lune
  - Research Site, Tauves
  - Research Site, Tence
  - Research Site, Thann
  - Research Site, Thenon
  - Research Site, Thilouze
  - Research Site, Thionville
  - Research Site, Thiviers
  - Research Site, Thoirette
  - Research Site, Thoré-la-Rochette
  - Research Site, Thouaré-sur-Loire
  - Research Site, Thun-Saint-Amand
  - Research Site, Thuré
  - Research Site, Tincques
  - Research Site, Torteron
  - Research Site, Toufflers
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tourrettes-sur-Loup
  - Research Site, Tours
  - Research Site, Traînel
  - Research Site, Trets
  - Research Site, Tréguier
  - Research Site, Troisfontaines
  - Research Site, Troissereux
  - Research Site, Turretot
  - Research Site, Ussac
  - Research Site, Ustaritz
  - Research Site, Uxem
  - Research Site, Uzès
  - Research Site, Vabres-l'Abbaye
  - Research Site, Vailly-sur-Aisne
  - Research Site, Vairé
  - Research Site, Valence-d'Albigeois
  - Research Site, Valenciennes
  - Research Site, Vals-les-Bains
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vannes
  - Research Site, Varennes-Vauzelles
  - Research Site, Veauche
  - Research Site, Vedène
  - Research Site, Vendeuil
  - Research Site, Verdelais
  - Research Site, Verdun
  - Research Site, Verfeil
  - Research Site, Vernet
  - Research Site, Versailles
  - Research Site, Vertus
  - Research Site, Vervins
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vénissieux
  - Research Site, Vézelise
  - Research Site, Vias
  - Research Site, Vic-en-Bigorre
  - Research Site, Vic-le-Comte
  - Research Site, Vienne
  - Research Site, Vif
  - Research Site, Vihiers
  - Research Site, Villaines-sous-Malicorne
  - Research Site, Villard
  - Research Site, Villard-Bonnot
  - Research Site, Ville-di-Pietrabugno
  - Research Site, Ville-la-Grand
  - Research Site, Villefranche-de-Lauragais
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villefranque
  - Research Site, Villelongue-de-la-Salanque
  - Research Site, Villeneuve-d'Ascq
  - Research Site, Villeneuve-Saint-Georges
  - Research Site, Villepinte
  - Research Site, Villers-Bretonneux
  - Research Site, Villers-Cotterêts
  - Research Site, Villers-Semeuse
  - Research Site, Villerupt
  - Research Site, Villette-d'Anthon
  - Research Site, Villiers-sur-Marne
  - Research Site, Violaines
  - Research Site, Vitré
  - Research Site, Vitrolles
  - Research Site, Vittel
  - Research Site, Vivier-au-Court
  - Research Site, Voinémont
  - Research Site, Voiron
  - Research Site, Vouillé
  - Research Site, Vrigne-aux-Bois
  - Research Site, Vœuil-et-Giget
  - Research Site, Wambrechies
  - Research Site, Wasselonne
  - Research Site, Wattignies
  - Research Site, Wattrelos
  - Research Site, Waziers
  - Research Site, Weitbruch
  - Research Site, Westhoffen
  - Research Site, Wignehies
  - Research Site, Wolfisheim
  - Research Site, Yerres
  - Research Site, Yerville
  - Research Site, Yvetot
  - Research Site, Yvré-l'Évêque